CLINICAL TRIAL: NCT06361862
Title: Does Continuous Vital Sign Monitoring Increase Investigations and Interventions in Complication-free Patients? - a Sub-study of Randomized Clinical Trials
Brief Title: Does Continuous Vital Sign Monitoring Increase Investigations and Interventions in Complication-free Patients?
Acronym: WARD-OT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Eske Kvanner Aasvang, Professor, head of research, MD, DmSci, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: WARD - Overtreatment
Record Dates: First submitted 2024-01-22; First posted 2024-04-12 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Cancer; Chronic Obstructive Pulmonary Disease; Surgery-Complications
MeSH Terms: conditions — Neoplasms; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- inactive alarms (No Intervention): Patients with continuous monitoring without active alerts from WARD.
- active alarms (Experimental): Patients with continuous monitoring with active alerts from WARD.
  Interventions: Device: Active alarms from WARD software

INTERVENTIONS:
Device: Active alarms from WARD software — Wireless continuous vital sign monitoring with real time staff alerts
  Arms: active alarms

SUMMARY:
This aim of this study is to investigate whether active alerts during CVSM result in an increased number of diagnostic tests and treatments in complication free patients, hypothesizing that more interventions are performed in the CVSM-group than standard of care (EWS) group.

ELIGIBILITY:
Inclusion Criteria:

* • Patients from WARD - RCT.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-04-02 (Actual); Study Completion 2025-04-02 (Actual)

PRIMARY OUTCOMES:
Frequency of patients having at least one of the following tests/treatments: | 72 hours
  * CT-scans
  * MRi-Scans
  * PET-Scans
  * X-ray (ordered by attending doctor, besides standard procedural investigations)
  * ultrasounds
  * Antibiotics (ordered by attending doctor, besides standard procedural treatment)
  * Arterial puncture
  * Gastro- colonoscopy
  * Dialysis
  * Central venous line (incl. dialysis catheter)

SECONDARY OUTCOMES:
The frequency of individual treatments and diagnostics: | 72 hours
  Treatments:
  * Antibiotics (ordered by attending doctor, besides standard procedural treatment)
  * CPAP
  * blood-transfusion
  * IV-fluids
  * Dialysis
  * Naso-gastric tube (ordered by attending doctor, besides standard procedural treatment)
  * Central venous line (incl. dialysis catheter)
  Diagnostics:
  * Imaging CT, X-ray, MRI, PET, and ultrasound.
  * Blood tests: arterial blood gases, cultures, and other blood sample tests.
  * ECG
  * cultures from urine, sputum, swabs, and feces.

CONTACTS AND LOCATIONS:
Locations (1):
- Eske Kvanner Aasvang, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No